CLINICAL TRIAL: NCT06499727
Title: HighCycle Study: Effect of Acetazolamide on Acute Mountain Sickness in Women Compared to Men: A Randomized, Placebo-Controlled, Double-Blind Parallel Trial
Brief Title: HighCycle Study: Effect of Acetazolamide on Acute Mountain Sickness in Women Compared to Men
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: National Center of Cardiology and Internal Medicine named after academician M.Mirrakhimov (Other Government); University Hospital Heidelberg (Other); Laboratoire des Adaptations Métaboliques à l'Exercice en conditions Physiologiques et Pathologiques (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HighCycle_AMS
Record Dates: First submitted 2024-07-05; First posted 2024-07-12 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-05

CONDITIONS: Acute Mountain Sickness
Keywords: Women; Hypoxia; Prevention; Acetazolamide; Altitude
MeSH Terms: conditions — Altitude Sickness; Hypoxia | interventions — Acetazolamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- WOMEN - ACETAZOLAMIDE oral capsule (Active Comparator): Acetazolamide 250 mg/day (capsules @125 mg; 1 in the morning, 1 in the evening), orally. Medication starts 24 hours before ascent to 3600 m until the morning after the second night at 3600 m.
  Interventions: Drug: Acetazolamide
- MEN - ACETAZOLAMIDE oral capsule (Active Comparator): Acetazolamide 250 mg/day (capsules @125 mg; 1 in the morning, 1 in the evening), orally. Medication starts 24 hours before ascent to 3600 m until the morning after the second night at 3600 m.
  Interventions: Drug: Acetazolamide
- WOMEN - PLACEBO oral capsule (Placebo Comparator): Placebo (capsules identically looking as acetazolamide capsules; 1 in the morning, 1 in the evening), orally. Medication starts 24 hours before ascent to 3600 m until the morning after the second night at 3600 m.
  Interventions: Drug: Placebo
- MEN - PLACEBO oral capsule (Placebo Comparator): Placebo (capsules identically looking as acetazolamide capsules; 1 in the morning, 1 in the evening), orally. Medication starts 24 hours before ascent to 3600 m until the morning after the second night at 3600 m.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetazolamide — Administration of 1x125mg acetazolamide in the morning, 1x125mg in the evening, starting 24 hours before departure to 3600 m.
  Arms: MEN - ACETAZOLAMIDE oral capsule; WOMEN - ACETAZOLAMIDE oral capsule
Drug: Placebo — Administration of equally looking placebo capsules in the morning and in the evening, starting 24 hours before departure to 3600 m.
  Arms: MEN - PLACEBO oral capsule; WOMEN - PLACEBO oral capsule

SUMMARY:
Millions of people travel to high altitude for work or leisure activities and are exposed to reduced inspiratory oxygen partial pressure and hypoxemia that may lead to altitude illness, among which the most common form is acute mountain sickness (AMS). The main AMS symptoms are headache, malaise, weakness, and fatigue. Prospective studies have shown that 20-60% of newcomers at 2500-4000m develop AMS requiring them to take medications, while, at very high altitudes, AMS may progress to high altitude cerebral oedema. Whether women are more susceptible to AMS remains insufficiently understood since no prospective study controlled for sex hormones, use of hormone contraception or assessed menstrual cycle phase (MCP) at altitude. Therefore, women remain underrepresented and poorly characterized in high altitude studies. In addition, the efficacy and safety of 250 mg/day acetazolamide, the standard recommendation for AMS prevention, has never been compared between sexes, although, women have presumably higher acetazolamide plasma concentration due to lower blood volume. Given the known dose-dependent preventive but also side effects of acetazolamide and equal proportion of women and men among mountain travellers, there is an urgent need to conclusively quantify the efficacy and safety of pre-ventive acetazolamide therapy against AMS in women compared to men.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking men and women, age 18-44 years, without any disease and need of regular medication (including oral contraceptives).
* BMI >18 kg/m2 and <30 kg/m2
* Born, raised and currently living at altitudes <1000 m
* Written informed consent
* Premenopausal women with an eumenorrheic cycle

Exclusion Criteria:

* Other types of contraceptvies (contraceptives (hormonal intrauterine device, vaginal ring, subcutaneous injections or implants, among others)
* Pregnancy or nursing
* Anaemic (haemoglobin concentration <10g/dl)
* Any altitude trip <4 weks before the study
* Allergy to acetazolamide and other sulfonamides

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 303 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Acute Mountain Sickness (AMS) Incidence, LLS 2018 | Day 1 to 3 at 3600 m
  Sex-related difference between acetazolamide and placebo group in the incidence of AMS. AMS incidence will be defined as a Lake Louise Questionnaire version 2018 score of ≥3.

SECONDARY OUTCOMES:
Acute Mountain Sickness (AMS) Incidence, LLS 1993 | Day 1 to 3 at 3600 m
  Sex-related difference between acetazolamide and placebo group in the incidence of AMS. AMS incidence will be defined as a Lake Louise Questionnaire version 1993 score of ≥3.
Acute Mountain Sickness (AMS) Severity, LLS 2018 | Day 1 to 3 at 3600 m
  Sex-related difference between acetazolamide and placebo group in the AMS severity assessed by the Lake Louise Questionnaire version 2018.
Acute Mountain Sickness (AMS) Severity, LLS 1993 | Day 1 to 3 at 3600 m
  Sex-related difference between acetazolamide and placebo group in the AMS severity assessed by the Lake Louise Questionnaire version 1993.
Drug-related side effects | Day 1 to 3 at 3600 m
  Sex-related difference between acetazolamide and placebo group in the incidence and severity of medication side effects.
Arterial blood gases | Day 2 at 760 m and day 2 at 3600 m
  Sex-related differences between acetazolamide and placebo group in the arterial blood gases (pH, PaO2, PaCO2, SaO2).
Acetazolamide plasma concentration | Day 2 at 3600 m
  Sex-related differences between acetazolamide plasma concentration assessed by dried blood spots.
Hypoxic ventilatory response | Day 2 at 760 m
  Sex-related difference in the hypoxic ventilatory response assessed under FiO2 of 0.115 and while cycling on a bicycle at 30% of predicted maximal work capacity.
Perceived pain visualization | Day 1 to 3 at 3600 m
  Sex-related differences between acetazolamide and placebo group on perceived pain sensations, visualized by the SMaRT tablet app

CONTACTS AND LOCATIONS:
Overall Officials: Michael Furian, Prof. Dr., Study Chair — University of Zurich; Talant Sooronbaev, Prof. Dr., Study Director — National Center of Cardiology and Internal Medicine, Bishkek, Kyrgyzstan
Locations (1):
- National Center for Cardiology and Internal Medicine, Bishkek, Gorod Bishkek, Kyrgyzstan

IPD SHARING:
Plan to Share IPD: Undecided